CLINICAL TRIAL: NCT02076061
Title: Biomarkers of Early Chronic Obstructive Pulmonary Disease (COPD) and Cardiovascular Diseases in Smokers/Ex-Smokers Attending Primary Care - Longitudinal Study
Brief Title: Biomarkers of Early Chronic Obstructive Pulmonary Disease (COPD) in Smokers - Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Örestadskliniken (Other)
Responsible Party: Principal Investigator, Johan Malm, Professor, Clincal Chemistry, Lund University
Other Study IDs: KOL 001
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Cardiovascular Disease; Lung Cancer
Keywords: COPD; Primary Care; Smoking; Smokers; ex-Smokers; Lung Cancer; Cardiovascular Disease; Proteomics; Biomarkers; Biobank; Disease Staging; Gold Stage
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Lung Neoplasms; Smoking; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- GOLD stage I
- GOLD Stage II
- GOLD Stage III
- GOLD Stage IV
- Smokers/ex-smokers w/o COPD
- non-Smokers w/o COPD

SUMMARY:
This is a longitudinal observational study to identify and validate protein biomarkers for COPD (chronic obstructive pulmonary diseases) and cardiovascular disease in smokers and ex-smokers attending primary care. Special emphasize is to correlate biomarkers to different phases of COPD, to progression of the disease, and to treatment of the disease. Furthermore, linkage between COPD, cardiovascular disease, and lung cancer will be investigated by identifying protein biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with COPD Gold stage 0-IV

Exclusion Criteria:

Patients with inflammatory diseases Patients with cancer Patients using immune system regulating drugs

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic in Malmö, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-02; Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Advanced disease etiology requiring hospitalization. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Johan Malm, Study Chair — Clincal Chemistry, Lund University; György Marko-Varga, Principal Investigator — Clinical Protein Science & Imaging, Lund University; Mikael Truedsson, Principal Investigator — Örestadskliniken Malmö; Elisabet Wieslander, Principal Investigator — Division of Oncology and Pathology, Lund University; Thomas E Fehniger, Principal Investigator — Clinical Protein Science & Imaging, Lund University; Magnus Dahlbäck, Principal Investigator — Clinical Protein Science & Imaging, Lund University; Roger Appelqvist, Principal Investigator — Clinical Protein Science & Imaging, Lund University
Locations (1):
- Örestadskliniken, Malmo, Sweden